CLINICAL TRIAL: NCT00365989
Title: A Clinical Study To Evaluate the Safety and Efficacy of MR Guided Focused Ultrasound Treatment of Uterine Fibroids With Enhanced Sonication Techniques
Brief Title: MR Guided Focused Ultrasound Treatment of Uterine Fibroids With Enhanced Sonication
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF018
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2018-12

CONDITIONS: Uterine Leiomyoma; Uterine Fibroids
Keywords: Fibroids; leiomyoma; neoplasm; benign tumors
MeSH Terms: conditions — Myofibroma; Leiomyoma; Neoplasms

ARMS (1):
- ExAblate Enhanced Sonication Test Arm (Experimental): The intervention to be administered is ExAblate Enhanced Sonication. The purpose of this study is to examine the safety profile of the ExAblate Enhanced Sonication mode to insure that no new safety issues are introduced compared to the normal focused ultrasound mode.
  Interventions: Device: ExAblate Enhanced Sonication

INTERVENTIONS:
Device: ExAblate Enhanced Sonication
  Other Names: Magnetic Resonance guided Focused Ultrasound

SUMMARY:
This is a phase 3 study to determine the safety of the new features to the FDA approved ExAblate device using a new method to ablate fibroids deemed Enhanced Sonication.

DETAILED DESCRIPTION:
Uterine leiomyoma (fibroids) are the most common neoplasms of the female pelvis. These benign tumors are generally oval in shape, and often highly vascular. On T2 weighted MR imaging exams, or T1 exams with contrast, uterine fibroids are easily identifiable. They occur in 20-25% of women of reproductive age and can cause a variety of problems generally described as either bleeding or mass effects from the fibroid. InSightec has developed an Enhanced Sonication (ES) technique for the ablation of these fibroids. This mode of tissue ablation has been added to the already FDA approved ExAblate system. The goal of this ES technique is to provide an additional treatment tool that will enhance the treatment effect without additional risks while preserving ALL clinical features of the current commercially approved version.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 18 or older, who present with symptomatic fibroids
2. Women who have given written informed consent
3. Women who are able and willing to attend all study visits.
4. Patient is pre or peri-menopausal (within 12 months of last menstrual period).
5. Able to communicate sensations during the ExAblate procedure.
6. Uterine fibroids, which are device accessible (i.e., positioned in the uterus such that they can be accessed without being shielded by bowel or bone).
7. Fibroids(s) clearly visible on non-contrast MRI.

Exclusion Criteria:

1. Women who are pregnant, as confirmed by serum test at time of screening, or urine pregnancy test on the day of treatment
2. Patient who desire to become pregnant in the future.
3. Patients who are breast-feeding.
4. Patients with an active pelvic inflammatory disease (PID)
5. Active local or systemic infection
6. Metallic implants that are incompatible with MRI
7. Known intolerance to the MRI contrast agent (e.g. Gadolinium or Magnevist)
8. Severe claustrophobia that would prevent completion of procedure in the MR unit.
9. Extensive abdominal scarring in the beam pass or dermoid cyst of the ovary anywhere in the treatment path.
10. Known or suspected pelvic carcinoma or pre-malignant conditions, including sarcoma and adenomatous hyperplasia.
11. Pedunculated fibroids.
12. Intrauterine device (IUD) anywhere in the treatment path
13. Undiagnosed vaginal bleeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Roberts, M.D., Principal Investigator — University of California, San Diego; Mark Shaman, M.D., Principal Investigator — KNI; Robert Min, M.D., Principal Investigator — Cornell; David Gianfelice, M.D., Principal Investigator — Toronto General Hospital; George Holland, M.D., Principal Investigator — Lahey Clinic
Locations (5):
- United States (4):
  - University of California at San Diego, La Jolla, California
  - Lahey Clinic, Burlington, Massachusetts
  - KNI, Kalamazoo, Michigan
  - Cornell Vascular, New York, New York
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- See also: Sponsor web page — http://www.insightec.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 83 subjects signing consent, 33 subjects failed additional study requirements and did not participate. Fifty (50) subjects were treated; 48 received enhanced sonications, 2 received only nominal sonications.
Groups:
- Enhanced Sonication Test Arm: ExAblate 2000 Enhanced Sonication (ES) mode generates higher ultrasound energy absorption at the focal volume compared to normal sonications.
Period: Overall Study
Arm/Group | Enhanced Sonication Test Arm
Started | 50
Completed | 48
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Population: Out of the 50 treated subjects, 48 received Enhanced Sonications (ITT) and 2 received only normal sonications.
Arm/Group | Enhanced Sonication Test Arm
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Only women with uterine fibroids qualified for this study.
  Participants
    Female | 48
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 11
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: The study objective is to determine the safety of the new Enhanced Sonication technique and assure no new safety issues are introduced.
Time Frame: Within 1 month of treatment
Measure: Number; unit: Adverse Events
Arm/Group | Enhanced Sonication Test Arm
Number analyzed (Participants) | 48
Adverse Events
  Total Adverse Events | 77
  Mild/Moderate Adverse Events | 75

2. Other Pre Specified Outcome: Mean Enhanced Sonication Normalized Thermal Dose Volume
Description: The secondary end point of the study is to evaluate the mean normalized Enhanced Sonication thermal dose volume. Normalized dose volume is a function of the sonication dose volume divided by the energy transmitted measured from the the MR thermometry imaging.
Time Frame: During treatment
Population: Of the 50 subjects treated, 39 were included in the thermal analysis per the protocol. Of the 11 subjects not eligible, 8 were not treated with at least 30% enhanced sonications. Three subjects received enhanced sonications at tissue depths greater that 70 mm from the skin line.
Measure: Mean (Standard Deviation); unit: cc/KJ/sonication
Arm/Group | Enhanced Sonication Test Arm
Number analyzed (Participants) | 39
cc/KJ/sonication | 0.67 (0.35)

3. Other Pre Specified Outcome: Number of Participants With Adverse Events
Time Frame: Within 1 month of treatment
Measure: Count of Participants; unit: Participants
Groups:
- ExAblate Enhanced Sonication Test Arm: The intervention to be administered is ExAblate Enhanced Sonication. The purpose of this study is to examine the safety profile of the ExAblate Enhanced Sonication mode to insure that no new safety issues are introduced compared to the normal focused ultrasound mode.
  ExAblate Enhanced Sonication
Arm/Group | ExAblate Enhanced Sonication Test Arm
Number analyzed (Participants) | 48
Participants
  Subjects with SAE reported | 0
  Subjects with no AEs reported | 13
  Subjects reporting AEs | 35
  Subject deaths | 0

ADVERSE EVENTS:
Arm/Group | Enhanced Sonication Test Arm
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 35/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Enhanced Sonication Test Arm (N=48)
All Pain/Discomfort (General disorders) | 32
Urinary tract infection (Renal and urinary disorders) | 5
Gastrointestinal (Gastrointestinal disorders) | 5
Abnormal Vaginal Discharge (Reproductive system and breast disorders) | 2/2
Skin burn (Skin and subcutaneous tissue disorders) | 1
Fever (General disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Migraine (Nervous system disorders) | 1
Dental (General disorders) | 1
Dizziness (General disorders) | 1
Edema (Skin and subcutaneous tissue disorders) | 1
IV bruise/numbness (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Heavy menses (Reproductive system and breast disorders) | 1
Abdominal cramping (Reproductive system and breast disorders) | 1
Leg pain - sonication related (Surgical and medical procedures) | 13
Abdominal pain - sonication related (Surgical and medical procedures) | 7
Back pain - sonication related (Surgical and medical procedures) | 7
Skin pain - sonication related (Surgical and medical procedures) | 6
Pain - sonication related (Surgical and medical procedures) | 2
Urinary frequency (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No